CLINICAL TRIAL: NCT00005023
Title: A Phase I Vaccine Trial of a HER-2/Neu Peptide Incorporated Into PLG Microspheres in Patients With Advanced Stage HER2-Expressing Cancers
Brief Title: Vaccine Therapy Plus Sargramostim in Treating Patients With Stage III or Stage IV Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Mary (Nora) Disis, Professor, University of Washington
Purpose: Treatment
Other Study IDs: CDR0000067339; UWASH-103; NCI-V99-1574
Record Dates: First submitted 2000-04-06; First posted 2004-04-23 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Lung Cancer; Ovarian Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage III non-small cell lung cancer; stage IIIB breast cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Adenocarcinoma of Lung | interventions — sargramostim

INTERVENTIONS:
Biological: HER-2/neu peptide vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to tumor cells. Colony-stimulating factors such as sargramostim increase the number of immune cells found in bone marrow or peripheral blood.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy plus sargramostim in treating patients who have stage III or stage IV cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of serial intradermal or subcutaneous vaccinations of HER-2 derived p369-377 peptide incorporated into polylactide-co-glycolide (PLG) microspheres with adjuvant sargramostim (GM-CSF) in patients with stage III or IV HER-2 expressing cancers. II. Determine whether cytotoxic T lymphocytes (CTL) specific for the HER-2 protein can be elicited in patients with HLA-A2 by immunization with this regimen. III. Determine which route of immunization, intradermal or subcutaneous, is more effective in generating HER-2 specific CTL in these patients on this regimen. IV. Determine the extent to which escalated dose of PLG peptide affects the immune response in these patients on this regimen.

OUTLINE: Patients undergo leukapheresis prior to study and after final vaccination. Patients are sequentially entered into one of three treatment arms: Arm I: Patients receive an intradermal vaccination of HER-2 derived p369-377 peptide incorporated into polylactide-co-glycolide (PLG) microspheres with adjuvant sargramostim (GM-CSF). Arm II: Patients receive a subcutaneous vaccination of HER-2 derived p369-377 peptide incorporated into PLG microspheres with adjuvant GM-CSF. Arm III: Patients receive a higher dose of subcutaneous vaccination of HER-2 derived p369-377 peptide incorporated into PLG microspheres with adjuvant GM-CSF. Treatment repeats every 4 weeks for up to 6 courses in the absence of unacceptable toxicity.

PROJECTED ACCRUAL: A total of 15 patients (5 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Stage III adenocarcinoma that overexpresses HER-2 and previously treated by surgical resection, conventional chemotherapy, or radiotherapy OR Stage IV adenocarcinoma that overexpresses HER-2 and in stable or complete remission with no other concurrent chemotherapy Must have documented HER-2 protein overexpression in the primary or metastatic tumor HLA-A2 positive

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 90-100% Life expectancy: At least 12 months Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Other: Female patients must have completed childbearing Fertile male patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior cytotoxic chemotherapy Endocrine therapy: At least 4 weeks since prior corticosteroids Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Other: No other concurrent investigational phase I studies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary (Nora) L. Disis, MD, Study Chair — University of Washington
Locations (1):
- University of Washington School of Medicine, Seattle, Washington, United States